CLINICAL TRIAL: NCT03511924
Title: Effect of Intradialytic Resistance Training on Circulatory miRNA Profile and Muscle Strength in Haemodialysis Patients
Brief Title: Intradialytic Resistance Training in Haemodialysis Patients
Acronym: IRTHEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pavol Jozef Safarik University (Other)
Collaborators: Dialysis Services Fresenius Medical Care Slovakia (Unknown); Private Health Institution Logman - Logman East (Unknown)
Responsible Party: Principal Investigator, Jaroslav Rosenberger, Jaroslav Resenberger, MD, PhD., Pavol Jozef Safarik University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PJSU-JR
Record Dates: First submitted 2018-04-13; First posted 2018-04-30 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: resistance training; circulating miRNA; muscle strength

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intradialytic resistance training (Experimental): During the 12-week intradialytic training plan subjects will be performed 3 to 5 sets of 3 different lower extremities exercises, each set will consist of 12 up to 18 repetitions of a single exercise. Subjects will take 1 to 2 minutes rest between each set. The resistance training will be realized 3 times per week and will be performed during haemodialysis therapy.
  Interventions: Behavioral: Intradialytic resistance training
- Control programme (No Intervention): Control subjects will receive no intervention during the 12-weeks of the experiment. Through the 12-week control period, all participants will be instructed to maintain a standard treatment regimen and to maintain their customary dietary and physical activity patterns.

INTERVENTIONS:
Behavioral: Intradialytic resistance training — Progressive resistance training programme performed during haemodialysis, taking into account subject´s medical review summarizing: A. full medical history, B. clinical examination including cardiovascular assessment, C. detailed medication usage history, D. review of recent biochemistry and haematology records and results of lower extremity muscle strength assessments. Construction of intradialytic training programme followed recommendations published by the Exercise & Sports Science Australia (Smart et al., 2013).
  Arms: Intradialytic resistance training

SUMMARY:
The study will investigate the effects of an intradialytic resistance training on miRNA´s expression and muscle strength in haemodialysis patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is accompanied by distortions of immune functions and acceleration of inflammation processes. Regular exercise has shown great potential for improving the health-related parameters of CKD patients. Moreover, muscle strength is considered to be an important predictor of protein- and energy- wasting, inflammation, quality of life and mortality in CKD patients. The behaviour and individual variability of adaptation to regular, controlled, supervised physical activities in CKD patients are not well defined and understood. The understanding of molecular adaptation mechanisms, represented by the epigenetic impact of exercise on renal specific miRNA´s expression, is necessary for future improvements in clinical practice. Monitoring pro- and anti-inflammation genes activity, their transcription factors and expression of miRNA molecules (influencing the signalling pathways of specific genes) will enable us to draft a new transcription and translation model for exercise-induced adaptation in CKD patients. Additionally, our results will indicate the clinical value of selected markers for the diagnostics and prognostics of disease.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 30 years of age, diagnosed with chronic kidney disease, treated with haemodialysis are eligible for our study.

Exclusion Criteria:

* Lower extremity amputation, severe dementia or retardation, acute intercurrent disease and probability of one year mortality higher than 25 % according to Charlson Comorbidity Index (CCI) are the exclusion criteria for participation in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-11 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Change in lower extremity muscle strength | Before the intervention, 1-5 days after the completion of the 12-week intervention and after 3 months follow up
  Change in maximal voluntary force produced during knee extension, leg flexion, extension and hip abduction, adduction will be assessed by dynamometer

SECONDARY OUTCOMES:
Change in activity of circulatory miRNA molecules involved in TRIM63 and IGF-1 signalling pathways | Before the intervention and 1-5 days after the completion of 12-week intervention
  Blood plasma will be collected for miRNAs analysis. We will analyze the activity of miRNAs involved in TRIM63 and IGF-1 signalling pathways for better definitions of chronic renal insufficiency and muscular adaptation following progressive resistance training. For miRNA analysis, we selected circulatory miRNA´s which were previously connected with regulation of calcium metabolism, calcification processes, protein-energy wasting, muscle mass and functions
Change in renal specific clinical data | Before the intervention, 1-5 days after the completion of the 12-week intervention and after 3 months follow up
  Clinical data will be collected from the medical documentation of patients. The extracted database will contain patient´s nephrological diagnosis profile, data about the presence of other diagnosis and comorbidities, body composition parameters and standard dialysis biochemistry, haematology and dialysis adequacy measures.
Change in score on the Hospital Anxiety and Depression Scale | Before the intervention and 1-5 days after the completion of 12-week intervention
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess states of depression and anxiety in the setting of a hospital medical outpatient clinic. The HADS consists of two subscales, subscale for anxiety and subscale for depression. Both subscales contains seven items and each item is rated on a four-point scale (numeric score range from 0 to 3 points). Maximal score for both subscales is 21, minimal score is 0. Scores of 11 or more on either subscale are considered to be a significant indicator of psychological morbidity. Scores between 8 and 10 represents "borderline" and scores between 0 and 7 represents "normal" indication of anxiety and depression.
Change in score on the Kidney Disease Quality of Life | Before the intervention and 1-5 days after the completion of 12-week intervention
  Kidney Disease Quality of Life (KDQOL™) instrument will be used to assess generic and kidney-disease targeted aspects of quality of life (self-rated health, self-rated change of health status, physical and mental component) of patients on haemodialysis.

OTHER OUTCOMES:
Satisfaction with Life Scale | 1-5 days before the intervention
  The Satisfaction With Life Scale will be used for measurements of the life satisfaction component of subjective well-being.
Multidimensional Scale of Perceived Social Support | 1-5 days before the intervention
  The Multidimensional Scale of Perceived Social Support will be used to measure how much support a parent feels they get from family, friends and significant others.
Health literacy | 1-5 days before the intervention
  The Health literacy level will be assessed using The Health Literacy Questionnaire and The Brief Health Literacy survey. This questionnaire comprises nine domains to provide a detailed profile of health literacy of populations, groups or patients of interest. The HLQ is divided into two parts which differ in response categories. Part 1 (domains 1-5) has 4 response categories rating the extent of agreement from 1 to 4. Part 2 (domains 6-9) has 5 response categories rating the level of difficulty from cannot do or always difficult (1), to always easy (5). Each domain was scored as the average of the item scores. The score ranges from 1 to 4 or 1 to 5 respectively, a higher score indicating higher level of health literacy.
Karnofsky Performance Status | 1-5 days before the intervention
  The Karnofsky Performance Status (KPS) scale will be used to assess self-sufficiency and functional capacity of patients on haemodialysis. KPS determines functional impairment in the performance of activities of daily living.
Subjective Global Assessment | 1-5 days before the intervention
  The nutritional status of patients will be assessed by Subjective Global Assessment method.

CONTACTS AND LOCATIONS:
Locations (1):
- Fresenius Medical Care - Dialysis Services Košice, Slovakia, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smart NA, Williams AD, Levinger I, Selig S, Howden E, Coombes JS, Fassett RG. Exercise & Sports Science Australia (ESSA) position statement on exercise and chronic kidney disease. J Sci Med Sport. 2013 Sep;16(5):406-11. doi: 10.1016/j.jsams.2013.01.005. Epub 2013 Feb 21. PMID 23434075
- [Derived] Zelko A, Rosenberger J, Kolarcik P, Madarasova Geckova A, van Dijk JP, Reijneveld SA. Age and sex differences in the effectiveness of intradialytic resistance training on muscle function. Sci Rep. 2023 Mar 1;13(1):3491. doi: 10.1038/s41598-023-30621-z. PMID 36859437